CLINICAL TRIAL: NCT04651101
Title: Can Vitamin D Deficiency be a Risk Factor of Coronary Artery Disease?
Brief Title: Vitamin D Deficiency in Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, Professor, Shiraz University of Medical Sciences
Other Study IDs: IR.SUMS.MED.REC.1398.246
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Coronary Disease
Keywords: coronary artery disease; vitamin D deficiency; Hs-CRP
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Vitamin D Deficiency | interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vitamin D deficient: those patient with vitamin D level below 30 ng/dl
  Interventions: Diagnostic Test: coronary angiography
- non vitamin D deficient: those patient with vitamin D above 30 ng/dl
  Interventions: Diagnostic Test: coronary angiography

INTERVENTIONS:
Diagnostic Test: coronary angiography — extent of coronary artery disease in invasive coronary angiography

SUMMARY:
Large population cross sectional study, was conducted between 2018-2020 by attendance of 4526 patients in shiraz, Iran. Patients were undergone selective coronary angiography from radial artery approach by an expert interventional cardiologist. 25-hydroxy vitamin D and Hs-CRP levels were measured for all patients

DETAILED DESCRIPTION:
This cross-sectional study was conducted in Shiraz. Clinical data were collected from the patients of Professor Kojuri cardiovascular clinic in Shiraz, Iran ( Iran, Fars Province, Shiraz, Niayesh Boulevard, Email: kojurij@yahoo.com, webpage: http://kojuriclinic.com/ )who came to clinic from March 2018 to March 2020. Inclusion criteria was all of the new patients who referred to Professor Kojuri cardiovascular clinic. Exclusion criteria were patients with more than 100ng/ml 25-hydroxy vitamin D3 serum level, parathyroid disorders, end-stage-renal-disease (ESRD) and paraneoplastic syndromes. Patients with more than 10mg/L Hs-CRP serum level also were excluded.

Complete history and physical exam were taken from the patients and risk factors such as hypertension, diabetes mellitus, age and gender were considered. 25-hydroxy vitamin D3 was checked for all patients. Blood pressure and took electrocardiography (ECG) for all patients were done. The dependent variable was the prevalence of Coronary Artery disease; the independent variable was vitamin D deficiency; and intervening factors were age, gender, hypertension, diabetes mellitus and level of Hs-CRP.

All Patients were undergone selective coronary angiography from radial artery approach by an expert interventional cardiologist. Angiography videos were reviewed by a team of expert cardiologists. Based on the results of coronary angiography, patients were classified as non-significant CAD with stenosis less than 50% and significant CAD with stenosis more than 50% stenosis. In this review diabetic and hypertensive patients is considered by criteria of American diabetes association 2018 & American heart association 2017 . Patient's serum level of 25-hydroxy vitamin D on their first visit was considered as index of vitamin D level. Vitamin D deficiency and sufficiency are defined respectively as serum level of 25-hydroxy vitamin D less than 30ng/ml and serum level of 25-hydroxy vitamin D more than 30 ng/ml . Patients with Parathyroid disorders and paraneoplastic syndromes were excluded

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected coronary artery disease who referred for coronary angiography

Exclusion Criteria:

* patients with Vitamin D more than 100ng/ml
* parathyroid disorders
* end-stage-renal-disease (ESRD)
* paraneoplastic syndromes
* Patients with more than 10mg/L Hs-CRP

Ages: 51 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: those who referred for coronary angiography with suspicion to coronary artery disease, who referred to our clinic
Sampling Method: Non-Probability Sample
Enrollment: 4526 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
coronary disease | 2 years
  extent of coronary artery disease in invasive coronary angiography
Hs-CRP | 2 years
  level of blood Hs-CRP as marker of inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Professor kojuri cardiology clinic, Shiraz, Outside of the US, Iran

IPD SHARING:
Plan to Share IPD: No
not distribute till publication